CLINICAL TRIAL: NCT05983497
Title: Effect of Self-care Skill Educational Intervention on the Compassionate Satisfaction and Compassionate Fatigue Among Clinical Nurses at HMC: A Randomized Controlled Trial
Brief Title: Effect of Self-care Skill Education on the Compassionate Satisfaction and Compassionate Fatigue Among Clinical Nurses Clinical Nurses at HMC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, Surekha Kiran Patil, Nurse Educator -II, Nursing and Midwifery Education Department, HMC, Principal Investigator, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MRC-01-22-581
Record Dates: First submitted 2023-07-25; First posted 2023-08-09 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Self-care; Compassion Satisfaction; Compassion Fatigue; Educational Intervention
MeSH Terms: conditions — Compassion Fatigue

STUDY DESIGN:
Intervention Model Description: This study uses a prospective, parallel group, randomized control group design to compare those received self-care skill educational intervention and the control group (no kind of intervention) among clinical nurses.
  The samples will be divided into experimental and control groups by randomly assigning the subjects to each group.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the study educational intervention, the subjects and investigators are not masked. However, the outcome assessors are marked for analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Self-care skill Education (Experimental): A total of 112 Participants will be assigned to the experimental group. Self-care skill educational intervention is administered to all the participants.
  Interventions: Other: Self-Care Skill Educational Intervention
- No Intervention: (No Intervention): A total of 112 Participants will be assigned to the control group.No intervention will be received

INTERVENTIONS:
Other: Self-Care Skill Educational Intervention — An evidence-based interactive self-care skill educational intervention that supports the clinical nurses to reduce compassion fatigue and increase the compassion satisfaction. The intervention will be delivered as 1-day activity-based educational training. The educational activity consists of the following content: the concept of compassionate fatigue, burnout awareness and recognition, eight dimensions of well-being, and followed by a demonstration of 7 guided self-care skill activities *on practicing sleep hygiene, self-talk, gratitude practice, Journaling, breathing exercise, heartfulness relaxation, and heartfulness meditation. After the activity participants will develop their own self-care plan for practicing the self-care skills. At the end of the session, they will receive the instructional leaflet to practice the 7 self care skills that they gained from the educational activity.
  Arms: Experimental: Self-care skill Education

SUMMARY:
The health of our nurses is perhaps the most important consideration for delivering excellent patient care. The passionate approach of nurses can lead to a lot of fatigue and stress among nurses. Their health is perhaps the most important consideration for delivering excellent patient care. Self-care provides nurses with the framework for managing professional burnout, compassion fatigue, and traumatic stress. The aim of this study is to assess the impact of self-care skill educational intervention on increasing compassion satisfaction and reducing compassionate fatigue among clinical nurses. The interactive Self-care skill education will be administrated and evaluated.

DETAILED DESCRIPTION:
Within the healthcare industry, healthcare professionals particularly nurses, are exposed to emotionally challenging and stressful situations, further, they experience increased levels of burnout and stress secondary to the nature of their work and work environment. The ability to manage work-related stress and burnout is vital to patient care and the individual health of nursing staff.

After the extensive literature search, it was identified that a dearth of studies was conducted in Qatar that explored the prevalence of burnout among different healthcare professionals. Most the of studies evaluated risk predictor and prevalence rate whereas no intervention studies to reduce the rates was found in Qatar. Organizational support through workplace intervention and the mitigating plan for the mental well-being of nurses is of utmost importance and has proven to be of merit. The researcher is interested to bring down the trend of the prevalence rate of compassionate fatigue through cost-effective self-care skill educational intervention among clinical nurses and to increase their compassionate satisfaction which in turn impacts nurses' work satisfaction and quality of care for patients.

The study aims to assess the effect of the self-care skill educational intervention on increasing compassion satisfaction among Nurses. This study uses a prospective, parallel group, randomized control group design to compare those who received Self -care Educational intervention to no intervention among clinical nurses. The samples will be divided into two groups and subjects will be randomly assigned to both groups. The research team will simple randomization method for randomly assigning the subjects to both arms.

A total of 224 samples are needed for the study. The samples will be randomly assigned to the two arms. The Professional Quality of Life Tool will be used for compassion fatigue and compassion satisfaction level among clinical nurses. This tool is considered valid and reliable. Assessment using ProQOL will be done at the beginning of administering the intervention and after 4 weeks of post-intervention.

An evidence-based interactive self-care skill educational intervention is developed by the research team and validated. The intervention will be delivered as 1-day activity-based educational training. The self-care skill educational intervention consist following content: the concept of compassion fatigue, burnout awareness and recognition, eight dimensions of well-being, concept of self-care and followed by a demonstration of 7 guided self-care skill activities sleep hygiene, self-talk, gratitude Practices, Journaling, breathing exercise, heartfulness relaxation, and heartfulness meditation. At the end of the educational intervention, Participants will receive an instructional leaflet to practice the 7 self-care skills that they gained from the educational activity. The participants are encouraged to practice based on the developed self-care plan.

The participants from the Control group will not receive any kind of intervention. after the 4 weeks assessed using ProQOL tool.

ELIGIBILITY:
Inclusion Criteria:

* Licensed registered Clinical nurses working all inpatient areas
* The nurses who are involved in direct patient care.
* Anticipated availability for the complete program.

Exclusion Criteria:

* New staff who are under preceptorship period.
* Clinical Nurses working in the outpatient department
* Staff who are not willing to participate

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 248 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2023-09-10 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Increase in the Compassion Satisfaction | 4 weeks
  The primary outcome will enhance the increase in compassionate satisfaction as assessed by using the ProQOL-5. The ProQOL tool is a standardized tool to assess compassion satisfaction and compassion fatigue which are valid and reliable.
  The ProQOL examines compassion satisfaction, burnout, and secondary traumatic stress. The 5-point Likert scale (1=Never to 5=Very often) is divided into 3 subscales of 30 items and 10 items measuring each concept. the Compassion satisfaction subscales range from 10- 50, the Higher score more than 23 indicates increase Compassion Satisfaction.
  The researcher is expecting an increase in compassion satisfaction levels among clinical nurses from the self-care skill educational intervention group as compared with non intervention group

CONTACTS AND LOCATIONS:
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No
All the data will be stored in a database by the principal investigator. Only PI will have access to the data base with a password. The Data will be shared only with the concerned research team member. The collected study data and analysis will be stored in the password-protected computer of the PI in NMED, HMC. The hard copies of the consent will be stored in a locker of P.I in NMED, HMC.
  Subject identifiers will not be shared outside HMC.